CLINICAL TRIAL: NCT05199025
Title: Biomarkers to Guide Perioperative Management and Improve Outcome in High-risk Surgery
Brief Title: Biomarkers in Perioperative Management
Acronym: BIGPROMISE
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, dr. P. Noordzij, Principal Investigator, St. Antonius Hospital
Other Study IDs: NL7407610020
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Complications; Quality of Life; Death
MeSH Terms: conditions — Postoperative Complications; Death | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Biomarker — Perioperative biomarker analyses

SUMMARY:
Rationale: The rate of postoperative complications after high-risk surgery remains high despite recent advances in perioperative management. There is a lack of objective and reliable information that can be used for risk stratification and to guide treatment decisions.

Objective: To describe the perioperative biomarker response in surgical patients with and without a postoperative complication and construct a preoperative and postoperative prediction model for postoperative complications. To systematically collect perioperative blood samples and clinical data in high-risk surgical patients for the development en analysis of biomarkers.

Study design: Multicenter, prospective, observational study. Study population: 4819 patients undergoing elective cardiac, colorectal, vascular and lung surgery.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: Main study parameters are levels of PCT, CRPhs, IL-6, GDF-15, sFLT, NT-proBNP, cTNThs, CysC and NGAL. Main study endpoint is the occurrence of a major postoperative complication which is defined as a surgical site infection, pneumonia, sepsis, acute kidney injury, major adverse cardiovascular events or death within 30 days of surgery.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In each patient five blood samples will be drawn for analysis. Most of the blood samples are drawn simultaneously with routine perioperative laboratory testing, which is common in this study population. In case a patient is admitted to the Intensive Care Unit blood samples will be collected using an arterial line. There are no direct risks or benefits for patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery (isolated coronary artery bypass grafting or combined with single valve surgery, isolated single valve surgery)
* Gastrointestinal surgery (colorectal, pancreatic, gastric surgery).
* Vascular surgery (open and endovascular aortic surgery, peripheral vascular surgery)
* Lung surgery (pneumonectomy,(bi)(sleeve)lobectomy or segmentectomy)

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Emergent surgery
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing surgery in the St. Antonius Hospital and the Amphia hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication | 30 days
  a surgical site infection, pneumonia, sepsis, acute kidney injury, major adverse cardiovascular events or death

SECONDARY OUTCOMES:
Failure to rescue | 30 days
  In-hospital death following a major complication
Mortality | 120 days
  Death
DAH120 | 120 days
  Days alive and out of hospital
Disability | 120 days
  Change in disability according to WHODAS 2.0 - 12 item

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amphia Hospital, Breda, North Brabant
  - St Antonius Hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Noordzij PG, Ruven HJ, Reniers T, Idema RN, Thio MS, Cremer OL, Hollema N, Smit KN, Vernooij LM, Dijkstra IM, Rettig TC. Cohort profile of BIGPROMISE: a perioperative biobank of a high-risk surgical population. BMJ Open. 2024 Jun 11;14(6):e078307. doi: 10.1136/bmjopen-2023-078307. PMID 38862228
- See also: Related Info — http://www.bigpromise.nl/ENG